CLINICAL TRIAL: NCT03552055
Title: Urine and Serum Concentrations of Pregnancy-Associated Compounds During Gestation
Status: Completed | Type: Observational
Sponsor: Gynuity Health Projects (Other)
Collaborators: University of Pennsylvania (Other); Planned Parenthood of Southeastern Pennsylvania (Unknown)
Responsible Party: Sponsor
Other Study IDs: 8000
Record Dates: First submitted 2017-04-20; First posted 2018-06-11 (Actual); Last update posted 2021-07-23 (Actual); Status verified 2021-07

CONDITIONS: Gestational Age
Keywords: placental proteins

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Biospecimen Retention: Samples With DNA — We will be collecting blood and urine specimens from participants for assay for five placental proteins.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Non-interventional Study — no interventions in this study, just specimen collection

SUMMARY:
Investigators will collect serum and urine specimens from pregnant patients along the full pregnancy continuum, assay each specimen for selected placental proteins, and examine the relationships between concentrations of the proteins and gestational age as determined by ultrasound.

DETAILED DESCRIPTION:
Investigators will collect serum and urine specimens from pregnant patients along with ultrasound results and information about factors that may affect the concentrations of proteins or the estimation of gestational age. Investigators will obtain data across the full pregnancy continuum but we will over sample patients within five gestational weeks before and after the 10 week mark.

Investigators will assay each specimen for selected placental proteins (Human placental lactogen (HPL), Schwangerschaftsprotein 1 (SP1), Pregnancy-associated plasma protein A (PAPP-A), A Disintegrin and Metalloproteinase 12 (ADAM12), and Human chorionic gonadotropin (HGC)) and any other proteins of interest identified prior to running assays and will examine the relationships between concentrations of the proteins and gestational age as determined by ultrasound.

The goal is to identify at least one compound and a concentration threshold for that compound that can be used for differentiating pregnancies of less than 10 weeks in duration from later pregnancies.

ELIGIBILITY:
Inclusion Criteria:

* Has an intrauterine pregnancy confirmed by ultrasound
* Not known to have pregnancy-induced hypertension (preeclampsia) or diabetes
* Not known to have a nonviable pregnancy, a multiple pregnancy, a pregnancy with a chromosomal or fetal abnormality, or a pregnancy with growth restriction
* Not currently taking anticoagulants
* Not currently having clinically significant vaginal bleeding, unusual pelvic pain, or other symptom suggestive of a pregnancy complication
* No use of assisted reproductive technology to conceive the current pregnancy
* Not previously enrolled in this study

Exclusion Criteria:

* Does not meet inclusion criteria

Sex: Female
Age Groups: Child, Adult, Older Adult
Study Population: Pregnant women
Sampling Method: Non-Probability Sample
Enrollment: 245 (Actual)
Dates: Start 2017-05-24 (Actual); Primary Completion 2018-03-30 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
protein concentration | 1 day
  Concentration of placental proteins in blood and urine

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Raymond, Principal Investigator — Gynuity Health Project
Locations (2):
- United States (2):
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Planned Parenthood of Southeastern Pennsylvania, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Raymond EG, Frye LJ, Weaver MA, Lebed JP, Ren X, Steider E, Winikoff B, Barnhart KT. Sensitivity and specificity of placental proteins for gestational age screening: An exploratory study. Contraception. 2020 May;101(5):309-314. doi: 10.1016/j.contraception.2020.01.007. Epub 2020 Feb 1. PMID 32014519